CLINICAL TRIAL: NCT07164534
Title: A Phase III Trial to Assess the Effectiveness of NRF2 Activator (Oral Sodium-copper- Chlophyllin ) in Locally Advanced Cervical Cancer to Reduce Late Radiotherapy Toxicity. (CHOC-LATE Trial)
Brief Title: A Clinical Trial to Assess the Effectiveness of NRF2 Activator (Oral Sodium-copper- Chlophyllin ) in Locally Advanced Cervical Cancer to Reduce Late Radiotherapy Toxicity.
Acronym: CHOC-LATE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Dr. Supriya Chopra, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4603
Record Dates: First submitted 2025-09-01; First posted 2025-09-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Uterine Cervical Neoplasm
Keywords: cervix cancer; radiation-related adverse effects; radiation; sodium-copper-chlorophyllin
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Chlorophyll

STUDY DESIGN:
Intervention Model Description: There will be Two Study Arm:
  If Patient Randomized to Arm 1 (Test arm) they will be given Oral adjuvant sodium-copper-chlorophyllin 750mg given once daily, on an empty stomach for 3 months, starting within 2 weeks of RT completion. If Patient Randomized to Arm 2 (Standard arm) they will receive Standard-of-care follow-up (no intervention) post RT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Test arm (Experimental): Oral adjuvant sodium-copper-chlorophyllin 750mg given once daily, given on an empty stomach for 3 months, starting within 2 weeks of radiotherapy completion
  Interventions: Dietary Supplement: Sodium-copper-chlorophyllin, a semi-synthetic derivative of chlorophyll, is made up of a mixture of sodium copper salts.
- Arm 2: Standard (No Intervention): Standard-of-care follow-up post radiotherapy

INTERVENTIONS:
Dietary Supplement: Sodium-copper-chlorophyllin, a semi-synthetic derivative of chlorophyll, is made up of a mixture of sodium copper salts. — Oral adjuvant sodium-copper-chlorophyllin 750mg given once daily given on an empty stomach for 3 months, starting within 2 weeks of RT completion
  Arms: Arm 1: Test arm

SUMMARY:
Cervical cancer is the second most common cancer in Indian women, and most patients are diagnosed at advanced stages.

The standard treatment for these stages is concurrent chemoradiotherapy, but this can cause long-term side effects such as bladder inflammation, strictures, ulcers, and tissue damage, which negatively impact patients' quality of life.

Previous studies have shown that oral sodium-copper-chlorophyllin can help reduce radiation-related side effects in rectal, prostate, and cervical cancer patients. However, no study has compared side effects between patients receiving standard follow-up care and those taking sodium-copper-chlorophyllin during follow-up.

We hypothesize that the use of sodium-copper-chlorophyllin as a short-duration adjuvant is associated with reduced incidence of late grade 2 or higher gastrointestinal and genitourinary toxicities compared to patients receiving standard-of-care follow-up.

DETAILED DESCRIPTION:
Descriptive summary

Objectives

Primary objective

• To assess the effectiveness of adjuvant sodium-copper-chlorophyllin in reducing the cumulative incidence of late grade 2 or higher RT-related gastrointestinal and genitourinary toxicity in cervix cancer patients, measured using the time-to-event method

Secondary objectives

* To evaluate the effect of sodium-copper-chlorophyllin tablet administration on 24-month local control, pelvic control, nodal relapse, disease-free survival, overall survival
* To compare the effect of sodium-copper-chlorophyllin on haematological parameters (persistent anaemia, neutropenia, thrombocytopenia)
* To compare the number of patients with RT-related urinary stress incontinence
* To examine the effect of diabetes mellitus, hypertension, bone health and vitamin deficiencies on the occurrence and recovery from RT-related toxicity
* To calculate cumulative time- and severity-related toxicity scores (C-MOSES scores)
* To compare prevalence of cystoscopic and sigmopidoscopy changes in test and standard arms and clinical symptoms in relation to the findings.
* To evaluate the quality of life in both arms
* To compare time spent in toxicity
* To calculate direct financial costs of adverse event management and impact on health care system.
* To investigate the effect of sodium-copper-chlorophyllin on the immune cell profile and oxidative stress markers of patients

Trial Design

This is a parallel-arm, randomized Phase III trial designed to test whether oral sodium-copper-chlorophyllin can reduce late (grade 2 or higher) gastrointestinal and genitourinary toxicities 24 months after completion of radiotherapy (RT) in cervical cancer patients.

Sample Size

Total of 316 patients will need to be randomized to the two arms in a 2:1 ratio (210 in the treatment group and 106 in the control group), accounting for an estimated 10%loss to follow-up. This sample size calculation was conducted using RPACT Package of R software.

Arm 1 (Test arm): Oral adjuvant sodium-copper-chlorophyllin 750mg given once daily, on an empty stomach for 3 months, starting within 2 weeks of RT completion

Arm 2 (Standard arm): Standard-of-care follow-up (no intervention) post RT

Patient will be selected as per Inclusion & Exclusion Criteria.

Inclusion criteria

* Female subjects aged 18 years or above with histologically proven locally advanced
* squamous cell or adenocarcinoma of the cervix
* Subjects eligible for RT and planned for definitive RT +/- chemotherapy with
* brachytherapy.
* Subjects who exceed the dose constraints of:

  * Rectum/sigmoid D2cm3 EQD23 by >70 Gy, or
  * Bladder D2cm3 EQD23 >80 Gy
* Subjects with adequate haematological, renal, hepatic and coagulation profiles and laboratory parameters within the following ranges:

  * Haemoglobin: ≥ 8 g/dl
  * ANC ≥ 1,500/mm^3
  * Platelet count 100,000/mm^3
  * Creatinine Clearance: ≥ 50 ml/min (as per Cockcroft-Gault formula)
  * Bilirubin: ≤ 2 x Upper limit of normal (ULN)
  * AST and ALT: ≤ 1.5 x ULN
* Subjects willing and able to comply with all study requirements, including treatment (e.g. able to swallow tablets), timing and/or nature of required assessments
* Ability to understand and willing to sign an informed consent document

Exclusion criteria

* Subjects with known hypersensitivity or contraindication to study drug or to any known component of study drug formulation
* Subjects with clinically significant decreased hematologic reserves, with major organ failure, severe electrolyte or metabolic abnormalities, any active infection or any other medical condition that may interfere with the ability to receive study treatment
* HIV positive patients
* Subjects with a history of blood dyscrasias
* Subjects consuming any other concurrent investigational agents
* Subjects with any other previous or current malignancy or RT that is likely to interfere with the protocol treatment or any other condition which according to the principal investigator might make an individual unsuitable for this study
* Subjects participating in any other clinical study within 90 days before enrolment in the study
* Subjects on active anti-coagulant treatment

Study Procedure

* All patients will have a baseline MRI or CT of the abdomen and pelvis.
* Concurrent chemoradiation and image-guided brachytherapy will be administered as per standard of care.
* Similarly, follow-up will be as per standard of care.
* During RT, patients will be evaluated weekly by investigators, and toxicities will be recorded using CTCAE v5.0 guidelines.
* Patients in the test arm will receive sodium-copper-chlorophyllin tablets (750 mg) once daily for 3 months, starting within 2 weeks of RT completion. Thus, a patient will take a total of 90 tablets. Sufficient tablets will be dispensed to the patient at each follow-up to last until the subsequent follow-up.
* Compliance to sodium-copper-chlorophyllin will be checked weekly by the study PI and study staff and through a patient drug logbook.
* The number of patients who do not complete the sodium-copper-chlorophyllin regimen will be noted, along with the reason for non-compliance.
* At the first follow-up, all patients will undergo clinical examination, blood collection and weight documentation.
* Radiological Examination will be done as per protocol.
* Patients will be followed post-completion of RT at 1 week for assessment of toxicity.
* Patients will be assessed at 3-month intervals for 2 years.
* for late grade ≥2 RT-related gastrointestinal and genitourinary toxicities and any other changes,
* Cystoscopies and sigmoidoscopies will be done.
* Cystoscopy and sigmoidoscopy will be performed twice a year for all patients.

Criteria for Adverse events

If there is suspicion of disease relapse, treatment will be given at the investigator's discretion.

Any grade 2 or higher nausea, vomiting or other sodium-copper-chlorophyllin-related adverse events will be reported in the case report forms. If any of the above adverse events lead to admission, serious adverse events (SAEs) will be reported to the IEC.

Statistical Plan

In this study, exploratory descriptive analyses and statistical analyses tests such as Kaplan-Meier, Chi-Square, Fisher's analysis and ANOVA will be conducted.

Baseline characteristics of patients in both study arms will be summarized using means and standard deviations for continuous variables and counts and percentages for categorical variables.

The primary efficacy endpoint will be assessed using Kaplan Meier Analysis using two-sided log rank test.

Secondary analyses will include logistic regression to adjust for confounders such as age and cancer stage with subgroup analyses based on HR-CTV and other relevant factors.

Time-to-toxicity will be evaluated using Kaplan-Meier survival analysis and log-rank tests for 2- and 3-year outcomes. Haematological parameters will be compared using Chi-Square or Fisher's exact tests.

Changes in Quality of Life (QOL) scores over a 2-year follow-up will be assessed using linear mixed modelling.

Average costs per grade of toxicity and according to arm of the study will be calculated. An Analysis of Variance (ANOVA) test will be considered to determine if there is a difference in costs between grades of toxicity, and an independent sample t-test will be used to determine if the average cost according to study arm is significantly different. The costs of study related additional cystoscopy and sigmoidoscopy are not included.

All analyses will be conducted using SPSS version 28, with a significance level set at 0.05.

Interim and full analyses will be performed.

Anticipated benefits of this study

If the trial results are positive, using adjuvant sodium-copper-chlorophyllin could potentially lower the incidence of late-grade toxicity associated with RT by 10% for cervical cancer.

This has the potential to improve the long-term quality of life for patients and reduce the costs associated with managing treatment-related side effects for both the healthcare system and patients.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged 18 years or above with histologically proven locally advanced squamous cell or adenocarcinoma of the cervix
* Subjects eligible for RT and planned for definitive RT +/- chemotherapy with brachytherapy.
* Subjects who exceed the dose constraints of:

  * Rectum/sigmoid D 2cm³ EQD2 ³ by more than 70 Gy, or
  * Bladder D 2cm³ EQD2 ³ more than 80 Gy
* Subjects with adequate haematological, renal, hepatic and coagulation profiles and laboratory parameters within the following ranges:

  * Haemoglobin: ≥ 8 g/dl
  * ANC ≥ 1,500/mm^3
  * Platelet count 100,000/mm^3
  * Creatinine Clearance: ≥ 50 ml/min (as per Cockcroft-Gault formula)
  * Bilirubin: ≤ 2 x Upper limit of normal (ULN)
  * AST and ALT: ≤ 1.5 x ULN
* Subjects willing and able to comply with all study requirements, including treatment (e.g. able to swallow tablets), timing and/or nature of required assessments
* Ability to understand and willingness to sign an informed consent document

Exclusion Criteria:

* Subjects with known hypersensitivity or contraindication to the study drug or to any known component of the study drug formulation
* Subjects with clinically significant decreased hematologic reserves, with major organ failure, severe electrolyte or metabolic abnormalities, any active infection or any other medical condition that may interfere with the ability to receive study treatment
* HIV positive patients
* Subjects with a history of blood dyscrasias
* Subjects consuming any other concurrent investigational agents
* Subjects with any other previous or current malignancy or RT that is likely to interfere with the protocol treatment, or any other condition which, according to the principal investigator, might make an individual unsuitable for this study
* Subjects participating in any other clinical study within 90 days before enrolment in the study
* Subjects on active anti-coagulant treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 316 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with cumulative late grade 2 or higher radiotherapy-related gastrointestinal and genitourinary toxicity incidence | 24 months
  Proportion of patients with cumulative late grade 2 or higher radiotherapy-related gastrointestinal and genitourinary toxicity incidence, reported using the time-to-event method, taken from the date of random assignment to the occurrence of late toxicity, or death because of late toxicity, at 24 months after completion of RT, by addition of sodium-copper-chlorophyllin for 3 months post RT (starting within 2 weeks of treatment completion), as compared to standard-of-care follow-up.

SECONDARY OUTCOMES:
Local Control at 24 months | 24 months
  Local Control: defined as the time interval between the date of random assignment and first evidence of local relapse.
Pelvic Control at 24 months | 24 months
  Pelvic Control: defined as the time interval between the dates of random assignment and first evidence of local and pelvic relapse
Nodal Relapse at 24 months | 24 months
  Nodal Control: defined as the time interval between the dates of random assignment and first evidence of any regional nodal relapse
Cumulative C-MOSES score | 24 months
  Cumulative time and severity incidence of toxicity scores (Months and Severity Score (MOSES) C-MOSES) for each patient, which is a toxicity summarising method that incorporates time
Proportion of patients with radiotherapy-related urinary stress incontinence | At treatment completion, 3 months, 6 months, 9 months
  Proportion of patients with RT-related urinary stress incontinence, as measured by the Oxford scale at treatment completion, 3 months, 6 months and 9 months after completion of RT
Disease-Free Survival at 24 months | 24 months
  Disease-Free Survival: defined as the time interval between date of random assignment and first relapse or death because of any cause.
Overall Survival at 24 months | 24 months
  Overall Survival: defined as the time interval between the date of random assignment and death due to any cause.
Proportion of patients with any acute toxicity | 4 weeks, 8 weeks and 12 weeks post radiotherapy completion
  Proportion of patients with any acute toxicity at treatment completion, 4 weeks, 8 weeks and 12 weeks after treatment completion.
Proportion of patients with any haematological abnormalities | 3 months and 6 months post radiotherapy completion
  Proportion of patients with any haematological abnormalities (anaemia, neutropenia, thrombocytopenia) at 3 months and 6 months after completion of RT
Patient-reported quality of life (QoL) | 3, 6, 9, 12, 15, 18, 21 and 24 months after radiotherapy completion
  Patient-reported quality of life (QoL) using EORTC-QLQ-C30 at baseline and all follow-ups
Cost of management of radiotherapy-related toxicity | 24 months
  Cost (in INR) of management of treatment-related toxicity in both arms

OTHER OUTCOMES:
Proportion of patients with comorbidities | At Day 1 and 24 Months
  Proportion of patients with pre-diabetes, diabetes mellitus and hypertension at baseline and follow-up
NRF2 levels | Day 1, After radiotherapy/before sodium-copper-chlorophyllin, 1 hour after sodium-copper-chlorophyllin, 3 hours after sodium-copper-chlorophyllin, 6 hours after sodium-copper-chlorophyllin
  Levels of NRF2 in all patients

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dasgupta A, Sawant S, Chatterjee A, Gota V, Sahu A, Choudhari A, Bhattacharya K, Puranik A, Dev I, Moiyadi A, Shetty P, Singh V, Menon N, Epari S, Sahay A, Shah A, Bano N, Shaikh F, Jirage A, Gupta T. Study Protocol of a Prospective Phase 2 Study of Chlorophyllin for the Management of Brain Radionecrosis in Patients With Diffuse Glioma (CHROME). Cancer Med. 2025 Mar;14(5):e70657. doi: 10.1002/cam4.70657. PMID 40025673
- [Background] Gagan Prakash DS, Supriya Chopra, Mahendra Pal, Amandeep Arora, Vedang Murthy, Lavanya Gurram, Prachi Mittal, Priyamvada Maitre, Mahendra Joshi, Shiv Madki, Sharath Kumar, Shraddha Bonkar Dethe, Priyal Gawad, Pankaj Chaturvedi, Tapan K Ghanty, Sudeep Gupta, Rajendra A. Badwe, Santosh Sandur, Vikram Gota. A phase II study of oral chlorophyllin in haemorrhagic cystitis secondary to radiation therapy for pelvic malignancies (CLARITY). 2024 ASCO Breakthrough; Yokohama, Japan. J Clin Oncol 42, 2024 (suppl 23; abstr 48): ASCO; 2024
- [Background] Egner PA, Munoz A, Kensler TW. Chemoprevention with chlorophyllin in individuals exposed to dietary aflatoxin. Mutat Res. 2003 Feb-Mar;523-524:209-16. doi: 10.1016/s0027-5107(02)00337-8. PMID 12628519
- [Background] Suryavanshi S, Sharma D, Checker R, Thoh M, Gota V, Sandur SK, Sainis KB. Amelioration of radiation-induced hematopoietic syndrome by an antioxidant chlorophyllin through increased stem cell activity and modulation of hematopoiesis. Free Radic Biol Med. 2015 Aug;85:56-70. doi: 10.1016/j.freeradbiomed.2015.04.007. Epub 2015 Apr 11. PMID 25872101
- [Background] Zhang Y, Guan L, Wang X, Wen T, Xing J, Zhao J. Protection of chlorophyllin against oxidative damage by inducing HO-1 and NQO1 expression mediated by PI3K/Akt and Nrf2. Free Radic Res. 2008 Apr;42(4):362-71. doi: 10.1080/10715760801993076. PMID 18404535
- [Background] Kumar SS, Shankar B, Sainis KB. Effect of chlorophyllin against oxidative stress in splenic lymphocytes in vitro and in vivo. Biochim Biophys Acta. 2004 May 3;1672(2):100-11. doi: 10.1016/j.bbagen.2004.03.002. PMID 15110092
- [Background] Park KK, Park JH, Jung YJ, Chung WY. Inhibitory effects of chlorophyllin, hemin and tetrakis(4-benzoic acid)porphyrin on oxidative DNA damage and mouse skin inflammation induced by 12-O-tetradecanoylphorbol-13-acetate as a possible anti-tumor promoting mechanism. Mutat Res. 2003 Dec 9;542(1-2):89-97. doi: 10.1016/j.mrgentox.2003.09.001. PMID 14644357
- [Background] Kumar SS, Devasagayam TP, Bhushan B, Verma NC. Scavenging of reactive oxygen species by chlorophyllin: an ESR study. Free Radic Res. 2001 Nov;35(5):563-74. doi: 10.1080/10715760100301571. PMID 11767414
- [Background] Stephens TJ, McCook JP, Herndon JH Jr. Pilot Study of Topical Copper Chlorophyllin Complex in Subjects With Facial Acne and Large Pores. J Drugs Dermatol. 2015 Jun;14(6):589-92. PMID 26091384
- [Background] Chernomorsky SA, Segelman AB. Biological activities of chlorophyll derivatives. N J Med. 1988 Aug;85(8):669-73. No abstract available. PMID 3050624
- [Background] Smith RG. Enzymatic debriding agents: an evaluation of the medical literature. Ostomy Wound Manage. 2008 Aug;54(8):16-34. PMID 18716339
- [Background] Dashwood RH. The importance of using pure chemicals in (anti) mutagenicity studies: chlorophyllin as a case in point. Mutat Res. 1997 Nov 28;381(2):283-6. doi: 10.1016/s0027-5107(97)00221-2. No abstract available. PMID 9434885
- [Background] Sudakin DL. Dietary aflatoxin exposure and chemoprevention of cancer: a clinical review. J Toxicol Clin Toxicol. 2003;41(2):195-204. doi: 10.1081/clt-120019137. PMID 12733859
- [Background] Chakraborty S, Mahantshetty U, Chopra S, Lewis S, Hande V, Gudi S, Krishnatry R, Engineer R, Shrivastava SK. Income generated by women treated with magnetic resonance imaging-based brachytherapy: A simulation study evaluating the macroeconomic benefits of implementing a high-end technology in a public sector healthcare setting. Brachytherapy. 2017 Sep-Oct;16(5):981-987. doi: 10.1016/j.brachy.2017.05.003. Epub 2017 Jun 7. PMID 28600140
- [Background] Jairam V, Lee V, Park HS, Thomas CR Jr, Melnick ER, Gross CP, Presley CJ, Adelson KB, Yu JB. Treatment-Related Complications of Systemic Therapy and Radiotherapy. JAMA Oncol. 2019 Jul 1;5(7):1028-1035. doi: 10.1001/jamaoncol.2019.0086. PMID 30946433
- [Background] Kirchheiner K, Potter R, Tanderup K, Lindegaard JC, Haie-Meder C, Petric P, Mahantshetty U, Jurgenliemk-Schulz IM, Rai B, Cooper R, Dorr W, Nout RA; EMBRACE Collaborative Group. Health-Related Quality of Life in Locally Advanced Cervical Cancer Patients After Definitive Chemoradiation Therapy Including Image Guided Adaptive Brachytherapy: An Analysis From the EMBRACE Study. Int J Radiat Oncol Biol Phys. 2016 Apr 1;94(5):1088-98. doi: 10.1016/j.ijrobp.2015.12.363. Epub 2015 Dec 29. PMID 26876955
- [Background] Vittrup AS, Tanderup K, Bentzen SM, Jensen NBK, Spampinato S, Fokdal LU, Lindegaard JC, Sturdza A, Schmid M, Segedin B, Jurgenliemk-Schulz IM, Bruheim K, Mahantshetty U, Haie-Meder C, Rai B, Cooper R, van der Steen-Banasik E, Sundset M, Huang F, Nout RA, Villafranca E, Van Limbergen E, Pieters BR, Tan LT, Lutgens LCHW, Hoskin P, Potter R, Kirchheiner K; EMBRACE Collaborative Group. Persistence of Late Substantial Patient-Reported Symptoms (LAPERS) After Radiochemotherapy Including Image Guided Adaptive Brachytherapy for Locally Advanced Cervical Cancer: A Report From the EMBRACE Study. Int J Radiat Oncol Biol Phys. 2021 Jan 1;109(1):161-173. doi: 10.1016/j.ijrobp.2020.08.044. Epub 2020 Aug 25. PMID 32853710
- [Background] Berveling MJ, Langendijk JA, Beukema JC, Mourits MJ, Reyners AK, Pras E. Health-related quality of life and late morbidity in concurrent chemoradiation and radiotherapy alone in patients with locally advanced cervical carcinoma. J Gynecol Oncol. 2011 Sep;22(3):152-60. doi: 10.3802/jgo.2011.22.3.152. Epub 2011 Sep 28. PMID 21998757
- [Background] Pras E, Willemse PH, Boonstra H, Hollema H, Heesters MA, Szabo BG, de Bruijn HW, Aalders JG, de Vries EG. Concurrent chemo- and radiotherapy in patients with locally advanced carcinoma of the cervix. Ann Oncol. 1996 Jul;7(5):511-6. doi: 10.1093/oxfordjournals.annonc.a010641. PMID 8839907
- [Background] Spampinato S, Fokdal LU, Potter R, Haie-Meder C, Lindegaard JC, Schmid MP, Sturdza A, Jurgenliemk-Schulz IM, Mahantshetty U, Segedin B, Bruheim K, Hoskin P, Rai B, Huang F, Cooper R, van der Steen-Banasik E, Van Limbergen E, Sundset M, Westerveld H, Nout RA, Jensen NBK, Kirisits C, Kirchheiner K, Tanderup K; EMBRACE Collaborative Group. Risk factors and dose-effects for bladder fistula, bleeding and cystitis after radiotherapy with imaged-guided adaptive brachytherapy for cervical cancer: An EMBRACE analysis. Radiother Oncol. 2021 May;158:312-320. doi: 10.1016/j.radonc.2021.01.019. Epub 2021 Feb 3. PMID 33545254
- [Background] Koom WS, Sohn DK, Kim JY, Kim JW, Shin KH, Yoon SM, Kim DY, Yoon M, Shin D, Park SY, Cho KH. Computed tomography-based high-dose-rate intracavitary brachytherapy for uterine cervical cancer: preliminary demonstration of correlation between dose-volume parameters and rectal mucosal changes observed by flexible sigmoidoscopy. Int J Radiat Oncol Biol Phys. 2007 Aug 1;68(5):1446-54. doi: 10.1016/j.ijrobp.2007.02.009. Epub 2007 May 7. PMID 17482766
- [Background] Trifiletti DM, Tyler Watkins W, Duska L, Libby BB, Showalter TN. Severe gastrointestinal complications in the era of image-guided high-dose-rate intracavitary brachytherapy for cervical cancer. Clin Ther. 2015 Jan 1;37(1):49-60. doi: 10.1016/j.clinthera.2014.11.003. Epub 2014 Nov 28. PMID 25444669
- [Background] Shejul J, Chopra S, Ranjan N, Mahantshetty U, Mehta S, Patil P, Engineer R, Gurram L, Phurailatpam R, Swamidas J, Gupta S, Shrivastava S. Temporal course of late rectal toxicity & impact of intervention in patients undergoing radiation for cervical cancer. Indian J Med Res. 2021 Aug;154(2):375-382. doi: 10.4103/ijmr.IJMR_4787_20. PMID 35142654
- [Background] Bologna E, Licari LC, Franco A, Ditonno F, Manfredi C, De Nunzio C, Antonelli A, De Sio M, Coogan C, Vourganti S, Leonardo C, Simone G, Autorino R. Incidence and Management of Radiation Cystitis After Pelvic Radiotherapy for Prostate Cancer: Analysis From a National Database. Urology. 2024 Sep;191:86-92. doi: 10.1016/j.urology.2024.04.035. Epub 2024 Apr 29. PMID 38692496
- [Background] Sturdza A, Potter R, Fokdal LU, Haie-Meder C, Tan LT, Mazeron R, Petric P, Segedin B, Jurgenliemk-Schulz IM, Nomden C, Gillham C, McArdle O, Van Limbergen E, Janssen H, Hoskin P, Lowe G, Tharavichitkul E, Villafranca E, Mahantshetty U, Georg P, Kirchheiner K, Kirisits C, Tanderup K, Lindegaard JC. Image guided brachytherapy in locally advanced cervical cancer: Improved pelvic control and survival in RetroEMBRACE, a multicenter cohort study. Radiother Oncol. 2016 Sep;120(3):428-433. doi: 10.1016/j.radonc.2016.03.011. Epub 2016 Apr 29. PMID 27134181
- [Background] Mazeron R, Fokdal LU, Kirchheiner K, Georg P, Jastaniyah N, Segedin B, Mahantshetty U, Hoskin P, Jurgenliemk-Schulz I, Kirisits C, Lindegaard JC, Dorr W, Haie-Meder C, Tanderup K, Potter R; EMBRACE collaborative group. Dose-volume effect relationships for late rectal morbidity in patients treated with chemoradiation and MRI-guided adaptive brachytherapy for locally advanced cervical cancer: Results from the prospective multicenter EMBRACE study. Radiother Oncol. 2016 Sep;120(3):412-419. doi: 10.1016/j.radonc.2016.06.006. Epub 2016 Jul 7. PMID 27396811
- [Background] Chopra S, Gupta S, Kannan S, Dora T, Engineer R, Mangaj A, Maheshwari A, Shylasree TS, Ghosh J, Paul SN, Phurailatpam R, Charnalia M, Alone M, Swamidas J, Mahantshetty U, Deodhar K, Kerkar R, Shrivastava SK. Late Toxicity After Adjuvant Conventional Radiation Versus Image-Guided Intensity-Modulated Radiotherapy for Cervical Cancer (PARCER): A Randomized Controlled Trial. J Clin Oncol. 2021 Nov 20;39(33):3682-3692. doi: 10.1200/JCO.20.02530. Epub 2021 Sep 10. PMID 34506246
- [Background] Kuku S, Fragkos C, McCormack M, Forbes A. Radiation-induced bowel injury: the impact of radiotherapy on survivorship after treatment for gynaecological cancers. Br J Cancer. 2013 Sep 17;109(6):1504-12. doi: 10.1038/bjc.2013.491. Epub 2013 Sep 3. PMID 24002603
- [Background] Spampinato S, Fokdal LU, Potter R, Haie-Meder C, Lindegaard JC, Schmid MP, Sturdza A, Jurgenliemk-Schulz IM, Mahantshetty U, Segedin B, Bruheim K, Hoskin P, Rai B, Huang F, Cooper R, van der Steen-Banasik E, Van Limbergen E, Sundset M, Westerveld H, Nout RA, Jensen NBK, Kirisits C, Kirchheiner K, Tanderup K; EMBRACE Collaborative Group. Importance of the ICRU bladder point dose on incidence and persistence of urinary frequency and incontinence in locally advanced cervical cancer: An EMBRACE analysis. Radiother Oncol. 2021 May;158:300-308. doi: 10.1016/j.radonc.2020.10.003. Epub 2020 Oct 14. PMID 33065183
- [Background] Georg P, Potter R, Georg D, Lang S, Dimopoulos JC, Sturdza AE, Berger D, Kirisits C, Dorr W. Dose effect relationship for late side effects of the rectum and urinary bladder in magnetic resonance image-guided adaptive cervix cancer brachytherapy. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):653-7. doi: 10.1016/j.ijrobp.2010.12.029. Epub 2011 Feb 23. PMID 21345618
- [Background] Spampinato S, Jensen NBK, Potter R, Fokdal LU, Chargari C, Lindegaard JC, Schmid MP, Sturdza A, Jurgenliemk-Schulz IM, Mahantshetty U, Hoskin P, Segedin B, Rai B, Bruheim K, Wiebe E, Van der Steen-Banasik E, Cooper R, Van Limbergen E, Sundset M, Pieters BR, Lutgens LCHW, Tan LT, Villafranca E, Smet S, Jastaniyah N, Nout RA, Kirisits C, Chopra S, Kirchheiner K, Tanderup K, Embrace Collaborative Group. Severity and Persistency of Late Gastrointestinal Morbidity in Locally Advanced Cervical Cancer: Lessons Learned From EMBRACE-I and Implications for the Future. Int J Radiat Oncol Biol Phys. 2022 Mar 1;112(3):681-693. doi: 10.1016/j.ijrobp.2021.09.055. Epub 2021 Oct 20. PMID 34678431
- [Background] Leiper K, Morris AI. Treatment of radiation proctitis. Clin Oncol (R Coll Radiol). 2007 Nov;19(9):724-9. doi: 10.1016/j.clon.2007.07.008. Epub 2007 Aug 28. PMID 17728120
- [Background] Potter R, Tanderup K, Schmid MP, Jurgenliemk-Schulz I, Haie-Meder C, Fokdal LU, Sturdza AE, Hoskin P, Mahantshetty U, Segedin B, Bruheim K, Huang F, Rai B, Cooper R, van der Steen-Banasik E, Van Limbergen E, Pieters BR, Tan LT, Nout RA, De Leeuw AAC, Ristl R, Petric P, Nesvacil N, Kirchheiner K, Kirisits C, Lindegaard JC; EMBRACE Collaborative Group. MRI-guided adaptive brachytherapy in locally advanced cervical cancer (EMBRACE-I): a multicentre prospective cohort study. Lancet Oncol. 2021 Apr;22(4):538-547. doi: 10.1016/S1470-2045(20)30753-1. PMID 33794207
- [Background] Gupta S, Maheshwari A, Parab P, Mahantshetty U, Hawaldar R, Sastri Chopra S, Kerkar R, Engineer R, Tongaonkar H, Ghosh J, Gulia S, Kumar N, Shylasree TS, Gawade R, Kembhavi Y, Gaikar M, Menon S, Thakur M, Shrivastava S, Badwe R. Neoadjuvant Chemotherapy Followed by Radical Surgery Versus Concomitant Chemotherapy and Radiotherapy in Patients With Stage IB2, IIA, or IIB Squamous Cervical Cancer: A Randomized Controlled Trial. J Clin Oncol. 2018 Jun 1;36(16):1548-1555. doi: 10.1200/JCO.2017.75.9985. Epub 2018 Feb 12. PMID 29432076
- [Background] Shrivastava S, Mahantshetty U, Engineer R, Chopra S, Hawaldar R, Hande V, Kerkar RA, Maheshwari A, Shylasree TS, Ghosh J, Bajpai J, Gurram L, Gulia S, Gupta S; Gynecologic Disease Management Group. Cisplatin Chemoradiotherapy vs Radiotherapy in FIGO Stage IIIB Squamous Cell Carcinoma of the Uterine Cervix: A Randomized Clinical Trial. JAMA Oncol. 2018 Apr 1;4(4):506-513. doi: 10.1001/jamaoncol.2017.5179. PMID 29423520
- [Background] Chopra S, Gupta M, Mathew A, Mahantshetty U, Engineer R, Lavanya G, Gupta S, Ghosh J, Thakur M, Deodhar K, Menon S, Rekhi B, Bajpai J, Gulia S, Maheshwari A, Kerkar R, Shylasree TS, Shrivastava SK. Locally advanced cervical cancer: A study of 5-year outcomes. Indian J Cancer. 2018 Jan-Mar;55(1):45-49. doi: 10.4103/ijc.IJC_428_17. PMID 30147092
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338